CLINICAL TRIAL: NCT04113460
Title: The Effectiveness Yoga@Work Among Office Workers With Chronic Nonspecific Neck Pain (CNNP): A Randomised Controlled Trial.
Brief Title: The Effectiveness Yoga@Work Among Office Workers With Chronic Nonspecific Neck Pain (CNNP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Yog-Kulam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMP/32491
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Chronic Non-Specific Neck Pain
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): The yoga group received the 8-week yoga sessions at work setting once a week by trained teacher followed by self practices.
  Interventions: Other: Yoga
- Control Group (No Intervention): Participants had one introductory session on proper physical position and stretching exercises to be practiced daily during work.

INTERVENTIONS:
Other: Yoga — Yoga@work program included physical movements, yoga posture, breathing exercise, pranayama and yoga chants. Session with trainer was conducted on worksite once a week for an hour.
  Arms: Yoga Group

SUMMARY:
Chronic nonspecific neck pain (CNNP) is a public health issues with a 50% life prevalence. CNNP is a leading cause of disability which contributes to higher costs due to loss of productivity, disability, and increased absenteeism from work. Yoga has been found effective managing neck pain but there has been no study at work setting for chronic non-specific neck pain.

To determine the effectiveness of Yoga@work program for chronic non specific neck pain among office workers, present randomised controlled trial was undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Participants who gave written informed consent
* Having neck pain for more than 3 month

Exclusion Criteria:

* Systematic disorder
* Neck or spine injuries
* Recent surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Neck Pain | Change from baseline to 8 weeks
  Pain was measured using Visual Analogue Scale

SECONDARY OUTCOMES:
Health related quality of life | Change from baseline to 8 weeks
  HRQoL was measured with the Short Form 36
Neck function | change from baseline to 8 weeks
  Neck functions with Northwick Park Neck Pain Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Yog-Kulam; Shekhar Sharma, Principal Investigator — NMP Medical Research Institute, India; Jaydeep Joshi, Study Chair — Yog-Kulam
Locations (1):
- Yog Bhawan, Jaipur, India

IPD SHARING:
Plan to Share IPD: Undecided